CLINICAL TRIAL: NCT01077206
Title: High-dose Simvastatin for Aneurysmal Subarachnoid Haemorrhage: Is it Better?
Brief Title: High-dose Simvastatin for Aneurysmal Subarachnoid Haemorrhage
Acronym: HDS-SAH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hong Kong Government (Other Government)
Responsible Party: Principal Investigator, George KC Wong, Professor (Clinical), Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GW005
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Aneurysm; statin; subarachnoid hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage; Aneurysm | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simvastatin 80mg (Active Comparator)
  Interventions: Drug: Simvastatin
- Simvastatin 40mg (Active Comparator)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — 80mg daily versus 40mg daily, for 21 days.
  Other Names: Teva

SUMMARY:
Experimental evidences supported the benefit of Simvastatin in subarachnoid haemorrhage. Moreover, Simvastatin is a potent agent in achieving low-density lipoprotein (LDL) reduction with a proven safety profile. However, there is no clinical data to compare the efficacy of different dosage regimens (namely whether high-dose regimen is better) and related cost-effectiveness analysis, although biochemical actions and related neuroprotective mechanisms were thought to be dosage-related. This gap in knowledge is important, on how to implement the use of statin and interpret different trial results. With these in mind, the investigators designed the current study.

Hypothesis:

Daily Simvastatin 80mg (high dose) treatment given within 96 hours of the ictus over three weeks will reduce incidence and duration of delayed ischemic deficits following subarachnoid haemorrhage when compared to daily Simvastatin 40mg (normal dose) treatment, leading to improvement in clinical outcome, which translates into advantage in terms of cost-effectiveness.

DETAILED DESCRIPTION:
Title: High-Dose Simvastatin for Aneurysmal Subarachnoid Haemorrhage (HDS-SAH): A multicentre randomised controlled double-blinded clinical trial.

Abstract

Background: Experimental evidence has indicated the benefit of simvastatin in the treatment of subarachnoid haemorrhage. Simvastatin is also a potent agent for reducing low-density lipoprotein (LDL). However, no clinical data are available to compare the efficacy of different dosage regimens (specifically, whether a high-dose regimen is more effective than a normal-dosage regimen) or conduct related cost-effectiveness analyses, even though the biochemical actions and related neuroprotective mechanisms are thought to be dosage-related. This gap in our knowledge of how to use statins and interpret trial results is very important, and motivated the investigators to conduct this study.

Objective: We hypothesized that eighty milligrams of simvastatin daily (high dose) over three weeks initiated within 96 hours of the ictus will reduce the incidence of delayed ischaemic deficits following subarachnoid haemorrhage when compared to 40mg of simvastatin daily (normal dose), leading to improvements in clinical outcomes and thus cost-effectiveness.

Methods: The study design is a randomised controlled double-blinded clinical trial (ClinicalTrials.gov Identifier: NCT01077206). Two hundred and forty aneurysmal subarachnoid haemorrhage patients (presenting within 96 hours of the ictus) from six neurosurgical centres are being recruited over three years. Primary outcome measure is Presence of delayed ischaemic deficits (DIDs). Secondary outcome measures include Modified Rankin Disability Score (mRS) at three months (favourable if 0-2) and Cost-Effectiveness Analysis in terms of overall direct cost per patient and incremental cost-effectiveness ratio (ICER).

Expected outcome: This will be the first study to clarify whether high-dose simvastatin is better than normal-dose simvastatin for patients with acute aneurysmal subarachnoid haemorrhage in terms of neurological outcomes and cost-effectiveness.

General Information

Protocol title: High-dose simvastatin for aneurysmal subarachnoid haemorrhage (HDS-SAH) ClinicalTrials.gov Identifier: NCT01077206 (Full protocol available online) Other Study ID Number: GW005 Name and address of the funding agency: Health and Health Service Research Fund (Reference Number: 07080401), Food and Health Bureau, Hong Kong Government, HKSAR, China Study protocol confirmed with grant funding body: 15 September 2009 Ethics approval of the study protocol: Joint CUHK-NTEC Clinical Research Ethics Committee, Hong Kong SAR, China

Study Investigators:

Steering Committee: Wong GK, Chan MT, Gin T, Siu DY, Leung MC Safety and data monitoring committee: Poon WS, Zee B Biostatistics: Zee B

Site investigators:

Department of Surgery, Prince of Wales Hospital, Hong Kong, China: Zhu XL, Wong GK; Department of Neurosurgery, the 8th Affiliated Hospital of Guangxi Medical University, Guangxi, China: M Liang; Department of Neurosurgery, Sichuan Province People's Hospital, Sichuan, China: HB Tan; Department of Neurosurgery, Pamela Youde Nethersole Eastern Hospital, Hong Kong, China: MW Lee, CK Wong; Department of Neurosurgery, Princess Margaret Hospital, Hong Kong China: TK Chan, YC Po; Department of Neurosurgery, Kwong Wah Hospital, Hong Kong China: PY Woo, KY Chan

Rationale and Background Information

Although aneurysmal subarachnoid haemorrhage (SAH) accounts for only 3-5% of strokes, its profound consequences and unique window of intervention justify its classification as a separate entity. Early aneurysm occlusion, expert endovascular neurosurgery and microsurgery, the use of oral nimodipine and neuro-intensive care are now the standards of care.1-3 Nevertheless, aneurysmal subarachnoid haemorrhage is still associated with mortality at one month for half of all patients, and the other half are left with disability.

Experimental evidence indicates the benefit of simvastatin in the treatment of subarachnoid haemorrhage.4-15 Simvastatin is also potent in reducing LDL, with a proven safety profile. Three randomised placebo-controlled pilot trials have supported the use of statins (two with 80mg of simvastatin and one with 40mg of pravastatin) for the treatment of aneurysmal subarachnoid haemorrhage.17-19 A systemic review has suggested that simvastatin may also reduce delayed cerebral ischaemia after aneurysmal subarachnoid haemorrhage,20 and another meta-analysis has recommended the routine use of statins in the care of patients with aneurysmal SAH.21 Finally, there is an ongoing multicentre, placebo-controlled phase III trial assessing the clinical benefits of treatment with 40mg of simvastatin daily [http://www.stashtrial.com/home.html].

However, no clinical data are available to compare the efficacy of different dosage regimens (specifically, whether a high-dose regimen is more effective than a normal-dosage regimen) or conduct related cost-effectiveness analyses, even though the biochemical actions and related neuroprotective mechanisms are thought to be dosage-related. This gap in our knowledge of how to use statins and interpret trial results is very important, and motivated the investigators to conduct this study.

Study Goal and Objective

The objective of the study is to determine whether a high dose of simvastatin for aneurysmal subarachnoid haemorrhage is superior to a normal dose in terms of clinical outcomes and cost-effectiveness. We hypothesized that eighty milligrams of simvastatin daily (high dose) over three weeks initiated within 96 hours of the ictus will reduce the incidence of delayed ischaemic deficits following subarachnoid haemorrhage when compared to 40mg of simvastatin daily (normal dose), leading to improvements in clinical outcomes and thus cost-effectiveness.

Study Design

The study design is a multicentre randomised controlled double-blinded (participants and outcome assessors) clinical trial.

Methodology

Subjects

Inclusion criteria:

1. Patients aged 18-70 years for whom the admitting neurosurgeon has a high index of suspicion of a spontaneous aneurysmal subarachnoid haemorrhage with convincing CT scan findings.
2. Any clinical grade, provided there is a reasonable prospect of survival.
3. The delay from the time of the presenting ictus until randomisation and the initiation of trial medication does not exceed 96 hours.

Exclusion criteria:

1. Unsalvageable patients: those with fixed and dilated pupils after resuscitation, and/or a devastating scan that preludes definitive therapy.
2. Previous statin therapy.
3. Current course of Warfarin-type drugs.
4. Pregnancy.
5. Known renal or hepatic impairment.
6. Suspected or known additional disease process that threatens life expectancy (e.g. malignancy).
7. Known or strong suspicion of drug abuse or alcoholism, or the likelihood of being amendable to either at the 3-month follow up.
8. Current course of amiodarone, verapamil or potent CYP3A4 inhibitors.

Outcome measures and follow-up:

Primary outcome measures:

1. Presence of delayed ischaemic deficits (DIDs): a fall of two or more points on the modified Glasgow Coma Scale, new focal neurological deficit lasting more than 2 hours, new cerebral infarction or CT perfusion evidence of cerebral ischaemia unrelated to surgery/embolisation, rebleed, hydrocephalus, infection, electrolyte or metabolic disturbance.

   Secondary outcome measures:
2. Modified Rankin Disability Score (mRS) at three months (favourable if 0-2).
3. Cost-effective analysis in terms of overall direct cost per patient and incremental cost-effectiveness ratio (ICER) of the high-dose group versus normal-dose group, i.e., the cost difference per patient divided by the difference in the percentage of (a) favourable outcomes and (b) delayed cerebral ischaemia. Sensitivity analyses for ICER will be carried out using the percentages of favourable outcomes and delayed cerebral ischaemia.

Study description

Ethical approval has been obtained from the respective institutional review boards. The study is adhering to the international quality standards provided in the Good Clinical Practice guidelines. After informed consent from patients or their next of kin, subjects are being randomised to receive 80mg of simvastatin (two tablets of 40mg each) or 40mg of simvastatin (one tablet of 40mg and one placebo tablet) per day for 21 days orally or through a nasogastric tube.

Randomisation Once the eligibility criteria have been fulfilled, a permuted-block randomisation is carried out using a computer system with an allocation list in random order generated by a statistician not related to the project team to protect the blinding and integrity of the study. The study drug assignments are concealed within sealed envelopes. These envelopes are only opened by site study investigators not involved in the clinical management of the recruited patients. The allocation ratio is 1:1. Both the clinical team (medical and nursing) and the patients are blinded to the study drug allocation.

Sample size Assuming that the high-dose group has a 35% delayed cerebral ischaemia risk with a 20% absolute reduction in delayed cerebral ischaemia as compared to the standard dose group with a 55% delayed cerebral ischaemia, a total of 212 patients will be required (80% power and 2-sided alpha=0.05). However, further assuming a 10% loss to follow up, 236 patients will need to be recruited. The study was designed with the expectation of 30 patients ¬being recruited at each of four centres per year22-23; a total of 240 patients is thus expected to be recruited over a 24 month period. Because of delays in starting patient recruitment in some centres, two extra centres (a total of six) were initiated for patient recruitment.

Trial status

Patient recruitment will be completed in March 2013, and the last recruited patient will be due for final outcome assessment in June 2013. Data archiving, data analyses and the dissemination of study results will take place in early 2014.

Safety Considerations

Drug-related morbidities including rhabdomyolysis and hepatitis have been rare. In the two reported pilot studies, only one patient withdrew due to elevated liver parenchymal enzymes, which reversed on cessation of medication. Plasma creatinine phosphokinase (CPK), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are being monitored for early signs of hepatitis or myositis every 7 days or on clinical suspicion. Administration of the study drug ceases if ALT/AST is more than three times the normal level of >180U/L or CPK >1,000U/L. Cholesterol levels are also monitored weekly.

Follow-Up

In addition to the laboratory tests mentioned above, the patients are followed up daily by the clinical team for any adverse events during acute admission and weekly for the first three weeks if discharged. A three-month clinical visit is arranged for outcome assessment and possible adverse event. A contact number is available for the enrolled patients for queries and suspected adverse event report.

Data Management and Statistical Analysis

Data are being collected on handwritten forms and archived in a password-protected electronic database.

We aim to perform an intention-to-treat analysis using two-sided probability, with P<0.05 considered statistically significant. Proportions with (a) DCI and (b) favourable outcomes will be compared with chi-square statistics. A sensitivity analysis for ICER will be carried out to find the limits of proportions of groups with (a) DCI and (b) favourable outcomes that show threshold values.

Planned exploratory analyses of DCI and favourable outcomes will include multivariate logistic regression using presentation SAH grade, age and the presence or absence of immediate post-procedural neurological deficits as the key covariates. Additional exploratory analyses with similar multivariate logistic regressions are planned, with the extra post-randomisation variables of the development of hydrocephalus, timing of hydrocephalus treatment and timing of aneurysm treatment.

Quality Assurance

The study conforms to the guideline of Good Clinical Practice. Data are managed in a secured computer system by a dedicated research assistants supervised by the principal investigator. The site investigators are contacted in case of doubt or uncertainty in data forms. The safety and data monitoring committee is being led by Professor Wai Sang Poon, Professor of Surgery, the Chinese University of Hong Kong. The committee is responsible for issues arising from the drugs used in the study, the interpretation of unexpected major adverse events, reviewing the study's progress and the submission of related recommendations to the study steering committee.

Expected Outcome of the Study

This will be the first study to clarify whether high-dose simvastatin is more effective than normal-dose simvastatin for patients with acute aneurysmal subarachnoid haemorrhage, in terms of neurological outcomes and cost-effectiveness. This gap in our knowledge of how to use statins and interpret trial results is very important.

Duration of Study

The initially targeted 24-month patient recruitment period has been extended to 30 months, with an additional 6 months required to complete the patient follow up and data archive. The total study period will thus be 36 months.

Project Management

The study steering committee is being led by the principal investigators. The committee is responsible for the study design, study implementation, ethics and health authority applications, protocol amendments, eventual data interpretation and the dissemination of results.

Statistical design and randomisation are being supervised by Professor Benny Zee, Division of Biostatistics, the Jockey Club School of Public Health and Primary Care, the Chinese University of Hong Kong.

The site study investigators are responsible for patient recruitment, reporting adverse events and completing the data collection.

Ethics

The study protocol was approved by the Joint CUHK-NTEC Clinical Research Ethics Committee, Hong Kong SAR, China. Ethical approval was obtained from the institutional review boards of the six neurosurgical centres. Written informed consent was obtained from eligible patients or next of kin for recruitment into the study.

References

1. Lovelock CE, Rinkel GJ, Rothwell PM. Time trends in outcome of subarachnoid hemorrhage: Population-based study and systemic review. Neurology. 2010; 74:1494-1501.
2. Wong GK, Ng RY, Poon WS. Aneurysmal subarachnoid haemorrhage. Surgical Practice. 2008; 12(2):51-55.
3. Wong GK, Boet R, Ng SC, Chan M, Gin T, Zee B, Poon WS. Ultra-early (within 24 hours) aneurysm treatment after subarachnoid hemorrhage. World Neurosurgery. 2012; 77:311-315.
4. Knuckey NW, Fox RA, Surveyor I, Stokes BA. Early cerebral blood flow and computerized tomography in predicting ischemia after cerebral aneurysm rupture. J Neurosurg. 1985; 62:850-855.
5. van Gijn J, Rinkel GJ. Subarachnoid haemorrhage: diagnosis, causes and management. Brain. 2001; 124:249-278.
6. STASH Trial. SimvaSTatin in Aneurysmal Subarachnoid Haemorrhage - a multicentre randomised controlled clinical phase III study protocol. www.stashtrial.com/Stash_pdf/2011/STASH%20study%20protocol.pdf.
7. Goldstein JL, Brown MS. Regulation of the mevalonate pathway. Nature. 1990; 343:425-430.
8. Delanty N, Vaughan CJ. Vascular effects of statins in stroke. Stroke. 1997; 28:2315-2320.
9. Vaughan CJ, Delanty N. Neuroprotective properties of statin in cerebral ischemia and stroke. Stroke. 1999; 30:1969-1973.
10. Wong GK, Poon WS. The biochemical basis of hydroxymethylglutaryl-CoA reductase inhibitors as neuroprotective agents in aneurysmal subarachnoid hemorrhage. Pharmaceuticals. 2010; 3:3186-3199.
11. Sabri M, Ai J, Marsden PA, Macdonald RL. Simvastatin re-couples dysfunctional endothelial nitric oxide synthase in experimental subarachnoid hemorrhage. PLoS ONE. 2011; 6:e17062.
12. Endres M, Laufs U, Huang Z, Nakamura T, Huang P, Moskowitz MA, Liao JK. Stroke protection by 3-hydroxy-3-methylglutaryl (HMG)-CoA reductase inhibitors mediated by endothelial nitric oxide synthase. Proc Natl Acad Sci. 1998; 95:8880-8885.
13. McGirt MJ, Lynch JR, Parra A, Sheng H, Pearlstein RD, Laskowitz DT, Pelligrino DA, Warner DS. Simvastatin increases endothelial nitric oxide synthase and ameliorates cerebral vasospasm resulting from subarachnoid haemorrhage. Stroke. 2002; 33:2950-2960.
14. Chen J, Zhang ZG, Li Y, Wang Y, Wang L, Jiang H, Zhang C, Lu M, Katakowski M, Feldkamp CS, Chopp M. Statin induce angiogenesis, neurogenesis, and synaptogenesis after stroke. Ann Neurol. 2003; 53:743-751.
15. Sugawara T, Ayer R, Jadhav V, Chen W, Tsubokawa T, Zhang JH. Simvastatin attenuation of cerebral vasospasm after subarachnoid hemorrhage in rats via increased phosphorylation of Akt and endothelial nitric oxide synthase. J Neurosci Res. 2008; 86:3635-3643.
16. Lynch JR, Wang H, McGirt MJ, Floyd J, Friedman AH, Coon AL, Blessing R, Alexander MJ, Graffagnino C, Warner DS, Laskowitz DT. Simvastatin reduces vasospasm after aneurysmal subarachnoid hemorrhage: results of a pilot randomized clinical trial. Stroke. 2005; 36:2024-2026.
17. Tseng MY, Czosnyka M, Richards H, Pickard JD, Kirkpatrick PJ. Effects of acute treatment with pravastatin on cerebral vasospasm, autoregulation, and delayed ischemic deficits after aneurysmal subarachnoid haemorrhage: a phase II randomized placebo-controlled trial. Stroke. 2005; 36:1627-1632.
18. Tseng MY, Hutchinson PJ, Czosnyka M, Richards H, Pickard JD, Kirkpatrick PJ. Effects of acute Pravstatin on intensity of rescue therapy, length of inpatient stay and 6-month outcome in patients after subarachnoid haemorrhage. Stroke. 2007; 38:1545-1550.
19. Chou SH, Smith EE, Badjatia N, Nogueira RG, Sims JR, Ogilvy CS, Rordorf GA, Ayata C. A randomized double-blind, placebo-controlled pilot study of Simvastatin in aneurysmal subarachnoid haemorrhage. Stroke. 2008; 39:2891-1893.
20. Tseng MY, the participants in the International Multidisciplinary Consensus Conference on the Critical Care Management of Subarachnoid Hemorrhage. Neurocrit Care. 2011; 15:298-301.
21. Sillberg VA, Wells GA, Perry JJ. Do statins improve outcomes and reduces the incidence of vasospasm after aneurysmal subarachnoid hemorrhage: a meta-analysis. Stroke. 2008; 39:2622-2626.
22. Wong GK, Chan TV, Poon WS, Boet R, Gin T. Intravenous Magnesium Sulphate to improve outcome after aneurysmal subarachnoid hemorrhage. Journal of Neurosurgical Anaesthesia. 2006; 18(2)142-148.
23. Wong GK, Poon WS, Chan MT, Boet R, Gin T, Ng SC, Zee BC. Intravenous magnesium sulphate for aneurysmal subarachnoid hemorrhage (IMASH): A randomized, double-blinded, placebo-controlled, multicenter Phase III Trial. Stroke. 2010; 41:921-926.

ELIGIBILITY:
Inclusion criteria:

1. Patients (age 18-70 years) in which the admitting neurosurgeon has a high index of suspicion of a spontaneous aneurysmal subarachnoid haemorrhage with a convincing CT scan findings.
2. Any clinical grade accepted provided a reasonable prospect of survival.
3. Delay to randomization and initiation of trial medication from the time of the presenting ictus does not exceed 96 hours.

Exclusion criteria:

1. Unsalvageable patients: Fixed and dilated pupils after resuscitation, and/or a devastating scan, which preludes definitive therapy.
2. Already taking statin therapy.
3. Those taking Warfarin-type drugs.
4. Pregnancy.
5. Known renal or hepatic impairment.
6. Suspected or known additional disease process, which threatens life expectancy (e.g. malignancy).
7. Known or strong suspicion of drug abuse, alcoholism, or those who are likely to be amendable to 3 month follow up.
8. Those already taking amiodarone, verapamil or potent CYP3A4 inhibitors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2010-09; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Presence of delayed ischemic neurological deficit | One month

SECONDARY OUTCOMES:
Liver function derangement or rhabdomyolysis | Three months
Modified Rankin Scale | Three months
Cost-effectiveness analysis | Three months

CONTACTS AND LOCATIONS:
Overall Officials: George KC Wong, Principal Investigator — Department of Surgery, The Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Wong GK, Chan DY, Siu DY, Zee BC, Poon WS, Chan MT, Gin T, Leung M; HDS-SAH Investigators. High-dose simvastatin for aneurysmal subarachnoid hemorrhage: multicenter randomized controlled double-blinded clinical trial. Stroke. 2015 Feb;46(2):382-8. doi: 10.1161/STROKEAHA.114.007006. Epub 2014 Dec 16. PMID 25516195
- [Derived] Wong GK, Liang M, Tan H, Lee MW, Po YC, Chan KY, Poon WS. High-dose simvastatin for aneurysmal subarachnoid hemorrhage: a multicenter, randomized, controlled, double-blind clinical trial protocol. Neurosurgery. 2013 May;72(5):840-4. doi: 10.1227/NEU.0b013e31828ab413. PMID 23392270